CLINICAL TRIAL: NCT02486601
Title: Phase II Study of NAB-PACLITAXEL Plus FOLFOX as Perioperative Chemotherapy in Patients With Operable Oesogastric Adenocarcinoma
Brief Title: NAB-PACLITAXEL Plus FOLFOX as Perioperative Chemotherapy in Patients With Operable Oesogastric Adenocarcinoma
Acronym: FOXAGAST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOXAGAST -D14-1
Record Dates: First submitted 2015-06-12; First posted 2015-07-01 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel + FOLFOX (Experimental): nab-paclitaxel + FOLFOX nab-paclitaxel: 150 mg/m2 D1 every 2 weeks Leucovorin: 400 mg/m2 D1 every 2 weeks Oxaliplatin: 85 mg/m2 D1 every 2 weeks 5-FU infusion: 2400mg/m2 48h infusion every 2 weeks 6 pre-operative cycles 6 post-operative cycles (optional)
  Interventions: Drug: nab-paclitaxel; Drug: FOLFOX

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel : 150 mg/m2 D1 every 2 weeks
  Other Names: ABRAXANE
Drug: FOLFOX — Leucovorin: 400 mg/m2 D1 every 2 weeks Oxaliplatin: 85 mg/m2 D1 every 2 weeks Fluorouracil (5-FU) infusion: 2400mg/m2 48h infusion every 2 weeks

SUMMARY:
This is a non-randomized pauci-centre, open-label phase II study. The treatment will consist in a chemotherapy by FOLFOX and nab-paclitaxel following modalities determined in the Brown University Phase I study.

In neoadjuvant setting : 3 months of treatment

Main criteria of Withdraw of the treatment: in case of tumor progression, non acceptable toxicity, or patient decision.

Post-operative treatment (for 6 additional cycles) is recommended, but will depend on the result of the neo-adjuvant treatment and the ability of patients to receive adjuvant chemotherapy based on tolerance of neo-adjuvant treatment and general post-operative condition (i.e. adjuvant treatment if no progression during neo-adjuvant chemotherapy, less than 80% of residual viable tumor compared to initial tumor volume, acceptable tolerance and post-operative PS 0 - 2). Adjuvant treatment must be initiated within 8 weeks post-operatively.

DETAILED DESCRIPTION:
This is a non-randomized pauci-centre, open-label phase II study. The treatment will consist in a chemotherapy by FOLFOX and nab-paclitaxel following modalities determined in the Brown University Phase I study.

In neoadjuvant setting : 3 months of treatment

Main criteria of Withdraw of the treatment: in case of tumor progression, non acceptable toxicity, or patient decision.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent, and willing and able to comply with protocol requirements,
* Histologically or cytologically proven adenocarcinoma of the low oesophagus or of the stomach, (from 1/3 inferior of the oesophagus to pylorus)
* HER2 negative tumors
* Localized and operable disease confirmed (stage I-III),
* No prior therapy for localized disease ,
* Age ≥18 years,
* Performance status (PS) 0-2,
* Haematological status: neutrophils (ANC) > 2.0x109/L; platelets >100x109/L; haemoglobin ≥9g/dL,
* Adequate renal function: serum creatinine level <150µM and creatinine clearance test > 30mL/min,
* Adequate liver function: AST (SGOT) and ALT (SGPT) ≤2.5xULN (Upper Limit of Normal)
* Total bilirubin ≤1.5 x ULN,
* Albumin ≥25g/L
* Baseline evaluations performed before inclusion: clinical and blood evaluations no more than 2 weeks (14 days) prior to inclusion, tumor assessment (CT-scan, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to inclusion,
* Female patients must be surgically sterile, or be postmenopausal, or must commit to using reliable and appropriate methods of contraception during the study and during at least six months after the end of study treatment (when applicable). All female patients with reproductive potential must have a negative pregnancy test (β HCG) within 72 hours days prior to starting nab-paclitaxel neo-adjuvant and adjuvant treatment. Breastfeeding is not allowed. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least six months after the end of the study treatment,
* Registration in a national health care system (CMU included for France).

Exclusion Criteria:

* Metastatic disease (stage IV)
* Non operable primary tumor
* Patient using warfarin,
* Uncontrolled hypercalcemia (corrected serum calcium > 2.55 mmol/l),
* Pre-existing permanent neuropathy (NCI grade ≥2),
* Known dihydropyrimidine dehydrogenase (DPD) deficiency,
* Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
* Treatment with any other investigational medicinal product within 28 days prior to study entry,
* Other serious and uncontrolled non-malignant disease (eg. active infection requiring systemic therapy, coronary stenting or myocardial infarction or stroke in the past 6 months),
* Known or historical active infection with HIV, or known active infection untreated with hepatitis B or hepatitis C.
* Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
* Patients with known allergy to any excipient of study drugs,
* Concomitant administration of live, attenuated virus vaccine such as yellow fever vaccine and concomitant administration of prophylactic phenytoin
* Patient with any medical or psychological condition, deemed by the investigator to likely interfere with patient's ability to sign informed consent or cooperate and participate in the study, including tutelage or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-10 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response rate | after three months of neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | time from the date of inclusion up to the date of disease progression or death whichever occurs last up to 7 years
Overall Survival (OS) | time interval form the inclusion to the date of the death from any cause up to 7 years
Health related to Quality of Life (QoL) | up to 8 months
Safety profile of the combination of nab-paclitaxel + FOLFOX regimen assessed by adverse events | time from randomisation up to end of study up to 7 years
Assessment of biomarkers when appropriate | 1 day of biopsie from diagnosis, and tumor from surgery
  such as SPARC, TS, DPD, ERCC1
Assessment of genetic polymorphism involved in tumor-response when appropriate | 28 days after last study treatment
  CYP2A6, TS, DPD, ERCC1, ERCC2

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LOUVET, Principal Investigator — Institut Mutualiste Montsouris
Locations (7):
- France (7):
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - CHU Pitie-Salpetriere, Paris
  - Hopital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris